CLINICAL TRIAL: NCT06240000
Title: Comparison of the Effectiveness of Radiofrequency Ablation of the Superior Cluneal Nerve and Conventional Physical Therapy in Patients With Chronic Low Back Pain
Brief Title: Radiofrequency Ablation of the Superior Cluneal Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Hüma Bölük Şenlikci, Associate Professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ankarasehir.kam@saglik.gov.tr
Record Dates: First submitted 2024-01-08; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Nerve Entrapment Syndrome; Radiofrequency Ablation; Low Back Pain
Keywords: Nerve Entrapment Syndrome; Radiofrequency Ablation; Low back pain
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Low Back Pain | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: This current prospective randomized study was carried out in Ankara Bilkent City Hospital, Department of Physical Therapy and Rehabilitation. Total of 25 CLBP patients (12 patients underwent SCN RFA, 13 patients participated CPT) were enrolled. Patients who admitted to outpatient clinics with low back pain that lasts more than 3 months, aged ≥ 18 year-old and detected positive 'iliac crest sign' included in the study. Patients have pain score <3 according to the Visual Analog Scale (VAS), INR >1.2 in blood samples were excluded from the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiofrequency ablation (Other)
  Interventions: Procedure: Radiofrequency ablation
- conventional physical therapy (No Intervention)

INTERVENTIONS:
Procedure: Radiofrequency ablation — Firstly, the posterior superior iliac spine was showed in the transverse plane, and it was gradually moved proximally until gluteus maximus muscle disappears and gluteus medius arises. Medial branch of the SCN is seen between iliac crest and thoracolumbar fascia as an ovoid structure. Radiofrequency device was utilized with 22-gauge 10-cm, 5 mm RF cannulas for all procedures. Cannula was placed thorough the SCN area and Sensory fiber stimulation was started between 0.3 and 0.5 V. The patient was asked for feedback on symptoms such as numbness, paresthesia or pain. If the patient did not report any sensory symptoms within the specified sensory stimulation range, the cannula was repositioned. Motor stimulation was given up to 1.5 V and it was checked whether there was any contraction or not. If there is no contraction detected, the SCN was ablated at 42° degrees centigrade for 240 seconds.
  Arms: Radiofrequency ablation

SUMMARY:
Low back pain is one of the most common musculoskeletal disorders affects individuals at least one during lifetime. Chronic low back pain (CLBP) lasts more than 3 months and decreases quality of life and causes work loss all over the world. Most common causes of Chronic Low back pain (CLBP) are lumbar disc herniation and/or degeneration, degenerative facet joints and sacroiliac joint pathologies, However, superior cluneal nerve (SCN) entrapment is another cause of CLBP that is ignored. It was reported that Superior cluneal nerve entrapment prevalence is % 1,6 - % 14 in CLBP patients. The Cluneal Nerves originate from the cutaneous branches of the dorsal ramus at T11-L4 and SCN innervates the skin of the upper part of the gluteal region. The nerves pass over the iliac crest through a tunnel formed by the thoracolumbar fascia and the upper edge of the iliac crest, that is the entrapment area. There are methods such as nerve blocks, neuromodulations and surgery in resistant cases. However, SCN entrapment is an overlooked diagnosis that should be considered in differential diagnosis.

Recently, radiofrequency ablation (RFA) of the SCN was performed under fluoroscopic guidance, total of 78% of patients reported nearly full analgesia for an average of 3 months. Although ultrasound-guided imaging and blocking of SCN is well described, there was not enough study that shows the effectiveness of ultrasound-guided SCN RFA and compares it to conventional physical therapy (CPT) in the treatment of CLBP.

ELIGIBILITY:
Inclusion Criteria:

1. Suffering from chronic low back pain more than 3 months
2. Age ≥ 18
3. VAS score ≥ 3/10
4. According to the blood samples, there should not be any detected bleeding diathesis (INR ≤1.2)
5. Patients detected positive 'iliac crest sign' included in the study

Exclusion Criteria:

1. Patients have pain score <3 according to the Visual Analog Scale (VAS)
2. INR >1.2 in blood samples
3. Radicular pain accompanying progressive neurological deficit
4. Sphincter disorder due to neurologic conditions
5. Local infections
6. Sepsis
7. Malignancy
8. Uncontrolled diabetes or other comorbidities leading general condition disorders
9. Allergic history related to used materials
10. Pregnancy
11. Mental disorders worsen cooperation were excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Visual analog Scale | Evaluated at baseline (pre-treatment), 2 weeks and 3 months after treatment completed
  Ten cm visual analog scale (VAS) was used by patients to perform a self-assessment of pain intensity associated with back pain. Higher scores indicate worse pain situations.

SECONDARY OUTCOMES:
Oswestry Disability Index | Evaluated at baseline (pre-treatment), 2 weeks and 3 months after treatment completed
  Index evaluating disability and functionality due to lumbar conditions consists of 10 self reported items. All questions are scored from 0-5. Higher scores indicates higher disability levels according to low back pain.
Short-Form 36 | Evaluated at baseline (pre-treatment), 2 weeks and 3 months after treatment completed
  The Short Form-36 (SF-36) is used to assess health related quality of life. The SF-36 consists of 36 items in mental and physical parts. Physical role, emotional role, physical function, energy/vitality, mental health, social function, pain, and general health are subgroups of the assessment. Scores range from 0 to 100, with higher scores indicating a better health-related quality of life. The Turkish validity and reliability of the SF-36 has previously been studied.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After writing is complete and submitted the journal, individual participant data is going to be shared
Supporting Information: Study Protocol, SAP
Time Frame: It will become available for 6 months after submitting

REFERENCES:
- [Result] Gautam S, Gupta N, Khuba S, Agarwal A, Kumar S, Das PK. Evaluation of the efficacy of Superior Cluneal Nerve Block in low back pain: A prospective observational study. J Bodyw Mov Ther. 2022 Apr;30:221-225. doi: 10.1016/j.jbmt.2022.03.001. Epub 2022 Mar 3. PMID 35500974
- [Result] Visnjevac O, Pastrak M, Ma F, Visnjevac T, Abd-Elsayed A. Radiofrequency Ablation of the Superior Cluneal Nerve: A Novel Minimally Invasive Approach Adopting Recent Anatomic and Neurosurgical Data. Pain Ther. 2022 Jun;11(2):655-665. doi: 10.1007/s40122-022-00385-x. Epub 2022 Apr 17. PMID 35430676
- [Result] Wu WT, Mezian K, Nanka O, Chen LR, Ricci V, Lin CP, Chang KV, Ozcakar L. Enhancing diagnosis and treatment of superior cluneal nerve entrapment: cadaveric, clinical, and ultrasonographic insights. Insights Imaging. 2023 Jul 3;14(1):116. doi: 10.1186/s13244-023-01463-0. PMID 37395948